CLINICAL TRIAL: NCT03024463
Title: The Multi-center Validation Study of Breast Cancer Internal Mammary Lymph Biopsy
Brief Title: The Multi-center Validation Study of Internal Mammary Lymph Biopsy With Modified Injection Technique in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Director of Breast Cancer Center, Shandong Cancer Hospital and Institute
Other Study IDs: IMLN-VS
Record Dates: First submitted 2017-01-09; First posted 2017-01-18 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Breast Neoplasm
Keywords: Breast Neoplasm; Internal Lymph Node; Sentinel Lymph Node Biospy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: IM-SLNB and IMLN dissection — Internal mammary sentinel lymph node biopsy followed by internal mammary lymph node dissection

SUMMARY:
In addition to axillary lymph node (ALN), internal mammary lymph node (IMLN) chain is also the first-echelon nodal drainage site for metastasis and it provides important prognostic information in breast cancer patients. However, decision about local treatment of IMLN is still being made based on ALN status. The 2016 National Comprehensive Cancer Network Guidelines recommend internal mammary lymph node irradiation for patients with more than 4 positive ALNs (category 1), and strongly consider irradiation for patients with 1 to 3 positive ALNs (category 2A). Therefore, there will be patients in positive ALN subgroup who just face complications of an unnecessary radiation to IMLN and there will be patients in negative ALN subgroup who do not receive adjuvant radiation therapy they really need. Thus, these inclusion criteria of National Comprehensive Cancer Network might lead to over-treatment and under-treatment. Internal mammary sentinel lymph node biopsy (IM-SLNB) provides a less invasive method of assessing the IMLN than surgical dissection. However, low visualization rate of IM-SLN has been a restriction of IM-SLNB. A modified radiotracer injection technique was established in our previous study. This technique could significantly improve the IM-SLN detection rate. The investigators have validated the accurate of the hypothesis and the modified radiotracer injection technique in the previous study.

For axillary sentinel lymph node biopsy, the success rate and the accuracy are the most important technical indicators. The relatively lower false-negative rate is a precondition for the widely application of SLNB. Axillary SLNB needs to be accomplished with the cooperation of multi-disciplinary teamwork, including the breast surgery, the radiologist, the nuclear medicine doctor and the pathologist, in order to obtain a better success rate and a lower false-negative rate. Our previous studies confirmed that the modified radiotracer injection technique can greatly improve the IM-SLN detection rate. However, whether the IM-SLNB based on the modified radiotracer injection technique has a low false negative rate or not still need to be confirmed by a further validation research.

Furthermore，recently, the investigators propose that if IM-SLN is the only metastatic lymph node and there would be no positive node else in IMLN chain, the radiotherapy and its associated complications could be avoided in these patients. On the other hand, if there is the presence of metastatic non-sentinel lymph node (NSLN) in IMLN chain after IM-SLNB, it is important to predict the risk of IM-NSLN metastasis in IM-SLN positive patients. As there is currently no such model, a predictive model for IM-SLN positive patients to avoid radiotherapy is needed in this situation. Therefore, a new study will be conducted to verify the issues above.

In the current study, all the participants (18~70 years of age) would have the preoperative pathology of invasive breast cancer and positive fine-needle aspiration result in their clinical or ultrasonic suspicious axillary lymph node. 99mTc-labeled sulfur colloid was injected into the parenchyma under the ultrasound guidance 3 to 18 hours before surgery. Two syringes of 9.25 to 18.5MBq 99mTc-labeled sulfur colloid in 0.5 to 0.7mL volume were injected at the 6 and 12 o'clock positions 0.5 to 1.0 cm from areola (about 2.0~4.0 cm from the nipple). IM-SLNB was performed in all participants with IMSLN visualized on preoperative lymphoscintigraphy and/or detected by the intra-operative gamma probe. All hotspots in the internal mammary basin were harvested and intra-operative identification of the IM-SLN was based on gamma probe detection. The IM-SLN was sectioned along the long axis into two blocks and all blocks were tested by the frozen section and the touch imprint cytology intra-operatively. Those participants with positive intra-operative results received IMLN dissection. Finally, all the IM-SLN blocks and IM-NSLN dissected were assessed post-operatively by H&E and Cytokeratin 19 stained immunohistochemistry. The conclusion would be drawn through the results mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Patients with preoperative pathology confirmed invasive breast cancer;
* Clinical N1-3 M0 (with positive fine-needle aspiration result in their clinical or ultrasonic suspicious axillary lymph node ; no clinical or radiologic evidence of distant metastases);
* Be able and willing to sign informed consent forms.

Exclusion Criteria:

* Patients who have received neoadjuvant therapy (including neoadjuvant chemotherapy and / or endocrine therapy);
* Patients with a previous history of breast cancer (recurrence of breast cancer and contralateral breast cancer);
* Patients with a history of other malignancies;
* Patients who have had previous surgery in axillary or internal mammary;
* Patients in pregnancy and lactation;
* Patients participant in other clinical trials that will have an impact on the results of this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 patients with positive axillary node
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
The accuracy (false negative rate) of internal mammary sentinel lymph node biopsy | Two years

SECONDARY OUTCOMES:
The number of internal mammary non-sentinel lymph node metastases in patients with positive axillary node and internal mammary sentinel lymph node | Two years
Factors influencing the number of internal mammary non-sentinel lymph node metastases in patients with positive axillary node and internal mammary sentinel lymph node | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China